CLINICAL TRIAL: NCT05235490
Title: Identification of Image Phenotypes to Predict Recurrence After Resection of Hepatocellular Carcinoma
Acronym: LIVERIBIOPSY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Median Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP191113
Record Dates: First submitted 2021-12-20; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: CT Scans Prior to Surgery With a Least 2 Years of Follow-up
Keywords: Hepatocellular Carcinoma; Hepatic resection; Biomarkers from CT scan; Prognostic value; Early recurrence with hepatocellular cancer patients
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non intervention — Data study with inclusion of patients and retrospective clinical data collection, combining :
  * Proofreading by radiologist of the CT scan performed (within 2 months prior to surgical intervention)
  * Proofreading by iBiopsy® of the CT scan performed (within 2 months prior to surgical intervention)
  * Proofreading of tumor sample slides by pathologists
  * Patients follow-up (imaging, clinical)
  * Recurrence-free survival

SUMMARY:
Tumor recurrence, which occurs in 70% of patients with HCC within 5 years after hepatic resection, is a major cause of post-resection-death. This recurrence can be true recurrence (intrahepatic metastases), which occurs sooner than 2 years later, or it can be due to the development of de-novo tumors at least 2 years later. Despite this high rate of tumor recurrence, no anti-recurrence adjuvant therapies are currently recommended.

Imaging phenomics is the systematic, large scale extraction of imaging features for the characterization and classification of disease phenotypes. Combining imaging and tissue phenomics could be a solution to predict HCC recurrence. With the emergence of molecular therapies and immunotherapies, identifying patients with HCC at high risk of post-resection recurrence would help determine additional therapeutic and management strategies in clinical practice.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is among the most lethal and prevalent cancers in the human population and it is now the third leading cause of cancer deaths worldwide, with over 500,000 people affected. Because of the high recurrence rate after curative hepatectomy, accurate prognostic assessment in HCC patients are quite important. With the emergence of molecular therapies and immunotherapies, the identification of patients at high or low risk for recurrence after hepatic resection would help determine additional therapeutic and management strategies in clinical practice. Although many immunohistochemical markers have been reported to have a prognostic value for HCC patients, there is no consensus on how these markers could add prognostic value to the clinical parameters.

In the initial step of biomarker discovery, no specific sample size is provided, however to test hypothesis, 100 patients are required.

This first study will potentially be followed by a second similar study promoted by the same investigators to increase the statistical power to improve the classification tool according to the patient's future.

Period covered by the data collection: 2011-2019 / Duration data collection: 1 year.

The primary endpoint will be built using machine learning method to obtain prediction of recurrence within 2 years. The Recurrence Free survival (RFS) within two years will be the reference outcome to evaluate the prognostic of the patients.

The secondary endpoint are following :

- A secondary endpoint which will be built using machine learning method to obtain prediction of recurrence after 2 years.

The Recurrence Free survival (RFS) after two years will be the reference outcome to evaluate the prognostic of the patients.

- A secondary endpoint will be the correlation between biomarker from CT scan and pathological biomarkers As the spectrum of HCC disease is very large, many patients to conduct conclusive validation studies for diagnostic and prognostic relevance need to be obtained.

Overall, each specific-read out endpoint will include a sample size calculation and - if appropriate - a power analysis specific to the objective of this study.

During training, phenotyping system performance assessment will be done to guide the calculation of the sample size for the validation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients who underwent surgery and have R0 resection after 2010
* Multiphase CT scans with contrast media should be performed within 2 months prior to surgical intervention
* At least 2 years of follow-up data on intrahepatic recurrence

Exclusion Criteria:

* Previous HCC treatment
* Combination of other anti-cancer treatment
* Other malignancies
* Patient expressly expressing opposition to the exploitation of their data as defined by the project
* Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients who has hepatectomy (resection R0) for an HCC treatment will be collected from January 2011 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
The main objective of this work is to identify biomarkers from CT scan (non-invasive imaging phenotypes from radiological images) which have a prognostic value for an early recurrence in patients with hepatocellular cancer. | 2 years
  The primary endpoint will be built using machine learning method to obtain prediction of recurrence within 2 years. The Recurrence Free survival (RFS) within two years will be the reference outcome to evaluate the prognostic of the patients.

SECONDARY OUTCOMES:
Identify biomarkers from CT scan (non-invasive imaging phenotypes from radiological images) which have a prognostic value for a tardive recurrence in patients with hepatocellular cancer. | 2 years
  A secondary endpoint which will be built using machine learning method to obtain prediction of recurrence after 2 years. The Recurrence Free survival (RFS) after two years will be the reference outcome to evaluate the prognostic of the patients.

OTHER OUTCOMES:
To correlate the imaging signatures predictive of recurrence with the cell population molding of tissue microenvironment (TME) and the tumor biology using tissue assessment as reference. | 1 year
  Correlation between biomarker from CT scan and nodule size, nodule differentiation (grade OMS), nodule capsule, macroscopie invasion, microscopic vascular invasion, macrotrabecular sub-type, satellite nodule, staging.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté LEWIN, Professor, Principal Investigator — Paul Brousse Hospital
Locations (1):
- Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: No